CLINICAL TRIAL: NCT05870787
Title: iMproving thE DIagnostics And Treatment Of ceRvical Precancer
Acronym: MEDIATOR
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0367531-3031
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2024-12

CONDITIONS: Cervical Dysplasia; Cervical Disease; Cervical Lesion; Cervical Cancer; Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Diseases; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Swede score colposcopy: Swede score colposcopy: includes application with acetic acid, supplemented with a systematic scoring system (the Swede score) including Lugols iodine, and collection of cervical biopsies.
  Interventions: Diagnostic Test: Swede score colposcopy
- Conventional colposcopy: Conventional colposcopy: includes application with acetic acid and collection of cervical biopsies.

INTERVENTIONS:
Diagnostic Test: Swede score colposcopy — New colposcopy method: with application of acetic acid, supplemented with a systematic scoringsystem (Swede score) including Lugols iodine, and collection of cervical biopsies.
  Groups: Swede score colposcopy

SUMMARY:
Cervical cancer screening is important as it enables identification of women at increased risk of the disease, but high-quality diagnostics of screen-positive women and effective treatment of those with precancer are critical in preventing progression to cancer. With the current transition from cytology-based to primary human papillomavirus (HPV)-screening and a growing proportion of HPV-vaccinated women, diagnostics of screen-positive women will become more challenging in the decades to come. Thus, there is a need to explore how to improve diagnostics while ensuring a low number of unnecessary procedures such as colposcopy and the collection of multiple cervical biopsies.

The overall purposes are:

Purpose 1: To investigate the diagnostic accuracy of cervical precancer when using a colposcopic scoring system in the diagnostic work-up of screen-positive women.

Purpose 2: To investigate the performance of a colposcopic scoring system to identify women without cervical precancer in whom collection of biopsies can be safely omitted.

DETAILED DESCRIPTION:
Introduction Cervical cancer is the fourth most common cancer in women worldwide. Every year, 375 women are diagnosed with cervical cancer in Denmark, and approximately 90 women die from the disease. Cervical cancer is caused by the sexually transmitted virus, human papillomavirus (HPV). When infected about 85-90 % clear the virus within a year or two. The remaining women develop a persistent HPV infection, which is associated with an increased risk of cervical intraepithelial neoplasia (CIN), which may progress to cancer if left untreated. Cervical cancer can be prevented through prophylactic HPV vaccination and screening. In Denmark, women aged 23 - 64 years are invited to the screening program. Women who do not participate in regular screening have an increased risk of cervical cancer, however up to 55% of cervical cancers are diagnosed in women who have attended screening. Hence, the performance of diagnostics is crucial.

Diagnostics Women with abnormal screening results may undergo repeat testing or be referred for colposcopy. Colposcopy allows the colposcopist to magnify and visualize the cervix with the transformation zone, where cervical cancer and cervical lesions typically arise. The aim is to make a colposcopic diagnosis and select the most severe area for biopsies, which undergo histopathological examination. Studies have shown considerable inter- and intra-observer variability even among experienced colposcopists, and a variable sensitivity of colposcopy as low as 55-57%. These findings suggest a need to improve the detection rate of CIN2+. A validated colposcopic scoring system, the Swede score, has been designed to improve the detection of high-grade cervical lesions, specified as cervical intraepithelial neoplasia grade 2 or worse (CIN2+) by providing an systematic approach to the colposcopy examination. The Swede score includes five variables (degree of 1) acetowhitening, 2) margins and surface, 3) vessels, 4) lesion size, and 5) iodine staining by using Lugols iodine) with a score from 0 - 2. Conventional colposcopy only utilizes acetic acid. In the original study, the Swede score had a high sensitivity and specificity for detecting high-grade cervical lesions (CIN2+), with an area under the receiver operating characteristics (ROC) curve of 0.87. Even so, the Swede score is endorsed by the International Agency for Research on Cancer (IARC/WHO) and by the European Federation for Colposcopy (EFC), it has not yet been implemented in Denmark. As previous studies have mostly evaluated the use of the Swede score among expert colposcopists, it is important to assess whether the score may be a valuable tool among non-experts. In Denmark, colposcopy is mostly performed by non-experts gynecologists. As a result of the low performance of colposcopy, and because several studies have shown that the CIN2+ detection rate increases with the number of biopsies collected, the Danish national guidelines recommend that all women should have a minimum of 4 biopsies collected. Biopsies should be collected from abnormal areas of the cervix and, if no lesion is detected, random biopsies should be taken. Our neighboring Scandinavian countries, for example Sweden and Finland, do not recommend collection of random biopsies. If biopsies could be omitted without increasing the risk of missing disease and reducing the harms with pain, bleeding and discomfort, this would benefit the women.

Aim

The project aims to explore whether the implementation of a systematic colposcopic scoring system, the Swede score, can:

Pupose 1: Improve diagnostic accuracy of cervical lesions with detection of CIN2+ in a Danish clinical setting.

Purpose 2: Evaluate whether the Swede score can be used to assess cervical lesions with <CIN1, so random biopsies can be safely omitted.

Data Characteristics of the women will be collected from medical records (previous gynecological historic, parity, smoking status, HPV-vaccination status, hormone use or immunosuppressive treatment). From the Danish Pathology Databank, we will collect data on previous screening history, result of the referral screening test, result of current and subsequent cervical biopsies and/or cervical excision.

ELIGIBILITY:
Inclusion Criteria:

* Women referred to colposcopy due to abnormal smear (HPV-genotype and cytology) in Central Denmark Region or Southern Denmark Region.

Exclusion Criteria:

* Allergic to iodine.
* Tranformationzone not visible (type 3).
* Atrophy of cervical epithelium.
* Women referred to colposcopy with no cervical biopsies taken or invalid cervical biopsies.
* Women with previous hysterectomy or without a cervix due to cervical cancer will be excluded.
* Pregnant women.

Ages: 23 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is focused on cervical cancer and precancer. Since only women have a cervix, only women will be included in this study.
Study Population: Women with abnormal smear (HPV-genotype and cytology) referred to colposcopy, visibel transformation zone (type 1 or 2) and where cervical biopsies has been sent to pathology examination.
Sampling Method: Non-Probability Sample
Enrollment: 929 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Purpose 1: Diagnosis of collected targeted cervical biopsies | When the histological report is available - typically within 12 weeks after the biopsy was taken
  The number of women diagnosed with Cervical Intraepithelial Neoplasia grade 2 or worse (CIN2+) diagnosed in cervical biopsies
Purpose 2: Diagnosis of collected random cervical biopsies | When the histological report is available - typically within 12 weeks after the biopsy was taken
  The number of women diagnosed with Cervical Intraepithelial Neoplasia grade 1 or less (<CIN1) vs. (CIN2+) diagnosed in random cervical biopsies.
  The clinical perspectives will be the absolute risk of CIN2+ in random biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hammer, MD, as.prof, Study Chair — University of Aarhus; Ulrik Schiøler Kesmodel, MD, prof, Study Chair — Aalborg University Hospital; Berit Bargum Booth, MD, Ph.d., Study Chair — Randers Regional Hospital; Line Winther Gustafson, MD, Ph.d., Study Chair — Aarhus University Hospital
Locations (7):
- Denmark (7):
  - Guldberg Kvindeklinik, Fredericia, Fredericia
  - Gødstrup Regional Hospital, Herning, Herning
  - Horsens Gynækologisk Klinik, Horsens, Horsens
  - Horsens Regional Hospital, Horsens, Horsens
  - Odense Univeristy Hospital, Odense, Odense
  - Randers Regional Hospital, Randers, Randers
  - Viborg Regional Hospital, Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knudsen AS, Randrup TH, Kesmodel US, Booth B, Gustafson L, Trope A, Strander B, Nieminen P, Hammer A. Assessment of a colposcopic scoring system (Swedescore) to reduce the number of cervical biopsies: a protocol for a clinical multicentre non-randomised intervention study in Denmark. BMJ Open. 2024 Dec 15;14(12):e085382. doi: 10.1136/bmjopen-2024-085382. PMID 39675832